CLINICAL TRIAL: NCT04533009
Title: Tramadol-paracetamol Combination in Treatment of Patients Undergoing Spinal Surgery
Acronym: TRAMAPARAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-11-10
Record Dates: First submitted 2018-05-04; First posted 2020-08-31 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo tablets are used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tramadol/acetaminophen (Active Comparator): Tramadol-paracetamol two tablets 37,5mg/325mg twice daily up to five days for patients undergoing spinal surgery
  Interventions: Procedure: spine surgery
- placebo (Placebo Comparator): Placebo two tablets twice daily up to five days for patients undergoing spinal surgery
  Interventions: Procedure: spine surgery

INTERVENTIONS:
Procedure: spine surgery — Tramadol-paracetamol 325mg/37,5mg two tablets twice daily

SUMMARY:
Tramadol-paracetamol combination is studied in patients coming for elective spine surgery. The study drug is started at the day of surgery and continued maximum of five days. Before the surgery pain, use of pain medication, satisfaction for pain medication, adverse effects, resilience, depression and life satisfaction were asked. At the discharge and seven days after the surgery use of pain medication and adverse effects were asked. The patients were followed up to 28 days and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years,
* BMI 18-35 kg/m2,
* informed consent obtained,
* elective spine surgery

Exclusion Criteria:

* Age<18 years or >75 years
* Hypersensitivity to anti-inflammatory drugs, paracetamol, tramadol or their auxiliary substances
* Acute or recovered hemorrhage in gastrointestinal tract or peptic ulcer
* Hemorrhagic disease
* Monoamineoxidase use in past two weeks
* Epilepsy
* Tendency to seizure
* Anti-seizure drugs in use Liver or renal failure Reduction in lung function Alcohol, drug or opioid addiction on record Acute intoxication due to alcohol, analgesics, opioids or psychopharmacon Pregnancy or breastfeeding Investigators estimation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction for pain medication | one week after surgery
  satisfaction measured with numeral rating scale 0-10 (0=not satisfied, 10= totally satisfied

SECONDARY OUTCOMES:
need for rescue pain medication | one week after surgery
  Measured as amount of other pain medicines used as rescue medicine
Pain assessment | one week after surgery
  Pain measered in numeral rating scale 0-10 (0= no pain, 10=worst pain)
adverse effects | one week after surgery
  Patient reported adverse reactions

OTHER OUTCOMES:
Pain assessment | one year after surgery
  Pain measered in numeral rating scale 0-10 (0= no pain, 10=worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No